CLINICAL TRIAL: NCT01996917
Title: Use of Prineo™ for Wound Closure in Breast Reduction Surgery
Brief Title: Use of Prineo in Breast Reduction Surgery
Acronym: Prineo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, Christine Hsu Rohde, MD, Assistant Professor of Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAM2053
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Efficiency of Surgical Incision Closure; Post-operative Scar
Keywords: wound closure; prineo; scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prineo closure (Active Comparator): One breast will have skin closure with Prineo.
  Interventions: Device: Prineo
- Standard Suture (No Intervention): One breast will be closed in the standard fashion with suture.

INTERVENTIONS:
Device: Prineo — After a Wise pattern breast reduction, one breast will have final layer closure with Prineo, while the other breast will be closed in the standard fashion with sutures.
  Other Names: Prineo wound closure system
  Arms: Prineo closure

SUMMARY:
This is a prospective, randomized, controlled, single-blinded study to compare Prineo™ with subcuticular sutures in 20 women undergoing bilateral breast reduction. For each patient, the final skin layer of one breast will be closed with subcuticular suture while the other breast will be closed with Prineo™. The treatment will be randomized to left or right breast. Therefore, the investigators will have 20 breasts in the suture group and 20 in the Prineo™ group, with each patient serving as her own control. For this study, the resident will close one side with suture and Dr. Rohde will apply the Prineo. The investigators will perform this study of incision closure under conditions as similar to normal conditions of closure.

DETAILED DESCRIPTION:
Wound closure with dermal sutures is time consuming and may increase risk of infection and inflammation. Moreover, appearance of the resulting scar depends largely on surgeon technique. Use of the Prineo™ wound closure system may decrease operative time, decrease incidence of infection and inflammation, and improve aesthetics of the resulting scar. Prineo™ has been shown to hold as well as sutures for the first 12-25 days and may reduce closure time of the final skin layer up to 75% in abdominoplasty and breast procedures. The system provides excellent coverage of the wound edge, protecting the incision with a microbial barrier. Cosmetic results in abdominoplasty and breast procedures appear to be equivalent to sutures.

The main endpoints will be operative time to closure of the final skin layer and patient-rated and blinded observer-rated scar quality. The investigators hypothesize that operative time to closure of the final skin layer using Prineo™ will be faster than operative time to closure using subcuticular suture. The investigators also hypothesize that subjective and objective scar quality of incisions closed with Prineo™ will be better than those closed with subcuticular suture.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing Wise pattern breast reductions for symptomatic macromastia.

Exclusion Criteria:

* Subjects who have an allergy to cyanoacrylate, formaldehyde, surgical tape, or any other known component of the Prineo system will be excluded.
* Subjects who refuse to be photographed or refuse to have their scars assessed by a blinded plastic surgeon will be excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rohde, MD,MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Dunst KM, Auboeck J, Zahel B, Raffier B, Huemer GM. Extensive allergic reaction to a new wound closure device (Prineo). Allergy. 2010 Jun 1;65(6):798-9. doi: 10.1111/j.1398-9995.2009.02243.x. Epub 2009 Nov 11. No abstract available. PMID 19909297

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 subjects were enrolled. Study procedures were performed per breast, therefore, each subject had one breast in the prineo arm and the other breast in the suture arm.
Units Other Than Participants: Breasts
Groups:
- Prineo Closure OR Standard Suture: One breast will have skin closure with Prineo.
  Prineo: After a Wise pattern breast reduction, one breast will have final layer closure with Prineo, while the other breast will be closed in the standard fashion with sutures.
  OR
  One breast will be closed in the standard fashion with suture.
Period: Overall Study
Arm/Group | Prineo Closure OR Standard Suture
Started | 21; 42 Breasts
Completed | 21; 42 Breasts
Not Completed | 0; 0 Breasts

BASELINE CHARACTERISTICS:
Population: 21 subjects were enrolled. Study procedures were performed per breast, therefore, each subject had one breast in the prineo arm and the other breast in the suture arm. The 21 subjects in the prineo arm are the same 21 subjects in the suture arm.
Units Other Than Participants: Breasts
Arm/Group | Prineo Closure OR Standard Suture
Number analyzed (Participants) | 21
Number analyzed (Breasts) | 42
Age, Continuous [Mean (Full Range); unit: years] | 37 [19 to 56]
Sex: Female, Male [Count of Participants; unit: Participants] — Only females were recruited for this study.
  Participants
    Female | 21
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 3
  More than one race | 0
  Unknown or Not Reported | 15
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Operative Time to Closure of Final Skin Layer
Description: This outcome measure looks at the operative time in seconds to closure of the final skin layer using Prineo or standard sutures.
Time Frame: During operation only
Population: 21 subjects were enrolled. Study procedures were performed per breast, therefore, each subject had one breast in the prineo arm and the other breast in the suture arm = a total 42 breasts.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Breasts
Arm/Group | Prineo Closure | Standard Suture
Number analyzed (Participants) | 21 | 21
Number analyzed (Breasts) | 21 | 21
seconds | 58.38 (2.11) | 444.76 (30.94)

2. Secondary Outcome: Score on Patient Observer Scar Assessment Scale (POSAS)
Description: The subject will complete the subjective part of the Patient Observer Scar Assessment Scale (POSAS) at each post-operative time point. Total score ranges from 6 to 60, with a higher score indicating a worse scar.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Breasts
Arm/Group | Prineo Closure | Standard Suture
Number analyzed (Participants) | 21 | 21
Number analyzed (Breasts) | 21 | 21
score on a scale
  2 Weeks | 30.5 (16.65) | 32 (15.98)
  1 Year | 25 (17.81) | 25.5 (18.39)

3. Other Pre Specified Outcome: Score on the Vancouver Scar Scale (VSS)
Description: A blinded plastic surgeon will evaluate objective scar quality using the Vancouver Scar Scale (VSS). Range of scores is from 0-13 with a higher score indicative of a worse scar.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Breasts
Arm/Group | Prineo Closure | Standard Suture
Number analyzed (Participants) | 21 | 21
Number analyzed (Breasts) | 21 | 21
score on a scale
  2 Weeks | 2.90 (1.47) | 4.1 (1.79)
  1 Year | 2.05 (1.04) | 2.2 (1.50)

ADVERSE EVENTS:
Arm/Group | Prineo Closure OR Standard Suture
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes